CLINICAL TRIAL: NCT04145765
Title: The Relationship of Risk Perceptions and Risk-taking With Humor Styles: Mediating Role of Self-control
Brief Title: Risk-taking, Self Control and Humor Styles
Status: Completed | Type: Observational
Sponsor: Malahat Amani (Other)
Responsible Party: Sponsor-Investigator, Malahat Amani, assistant professor, University of Bojnord
Organization: University of Bojnord (Other)
Other Study IDs: 13181
Record Dates: First submitted 2019-10-24; First posted 2019-10-31 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Risk-Taking; Humor as Topic; Self-Control
MeSH Terms: conditions — Risk-Taking; Self-Control

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: correlation — the subjects completed the questionnaires
  Other Names: descriptive

SUMMARY:
Therefore, this study tries to examine relationships among risk perception, risk-taking and humor styles through the mediating role of self-control. The present study used the correlation method. The statistical population consisted of all undergraduate students from University of Bojnord. The number of 400 students from the Faculty of Humanities and Basic Sciences was selected by using cluster sampling. The questionnaires were distributed in the classes among who inclined to participate in this study and they completed the questionnaires as anonymous.

ELIGIBILITY:
Inclusion Criteria:

* be a student of the college

Exclusion Criteria:

* Unwillingness to study And not being a student at university

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The numbers of 380 completed questionnaires were collected. The participants were in range 18 to 29 years old and the mean and standard deviation were 20.27 and 1.96, respectively. Given at the University of Bojnord the proportion of females to males is 70 percent to 30 percent that the proportion of females and males in the sample was observed. In this manner, the 78 percent, 17.7 percent and 4.4 percent of participants were female, male and uncertain, respectively.
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Self-Control | 2 days
  variable self-control was measured by the self-control Questionnaire. it has 36 items that were rated on a 5-point scale (from 1 not at all like me to 5 very much like me). it was completed by the participants.
Humor styles | 2 days
  variable of humor style was measured by the Questionnaire of humor style. it HSQ included 32-item measures humor styles on a 7-point Likert scale ranging from "strongly disagree (1)"to "strongly agree(7)". HSQ measure the four humor styles of affiliative, self-enhancing, aggressive, and self-defeating. it was completed by the participants.
risk taking | 2 days
  the variable of risk-taking was measeured by Domain-Specific Risk-Taking (DOSPERT) scale. DOSPERT is 30- items that measure risks in 5 fields: health/safety, social, ethical, financial, and recreational. Each item is assessed twice, one time was rated items based on perceived risk and next time was rated same items based on likelihood engage in the risky. it was completed by the participants.
  Responses are give with using a 7-point rating scale ranging from1 (Extremely Unlikely) to 7 (Extremely Likely). Higher scores indicate greater risk taking in the domain of the subscale.
  the risk-perception scale evaluates the respondents' gut level assessment of how risky each behavior is on a7-point rating scale ranging from 1 (Not at all) to 7 (Extremely Risky). Ratings are again added across all items of a given subscale to obtain subscale scores, with higher scores suggesting perceptions of greater risk in the domain of the subscale

CONTACTS AND LOCATIONS:
Overall Officials: Malahat Amani, Principal Investigator — University of Bojnord
Locations (1):
- university of Bojnord, Bojnourd, North Khorasan, Iran